CLINICAL TRIAL: NCT00049413
Title: Pentostatin, Cyclophosphamide And Rituximab (PCR) For B-Cell Chronic Lymphocytic Leukemia (CLL) And Small B-Cell Lymphocytic Lymphoma (SLL): Four Phase II Trials With Patient Stratification Based On Prior Therapy
Brief Title: Combination Chemotherapy and Rituximab in Treating Patients With Chronic Lymphocytic Leukemia or Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Cancer Biotherapy Research Group (Other)
Responsible Party: Robert O. Dillman, MD, Hoag Memorial Hospital Presbyterian
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258096; CBRG-NIP-0201; NCI-V02-1712; SUPEREN-CBRG-NIP-0201
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Leukemia; Lymphoma
Keywords: B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent small lymphocytic lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cyclophosphamide; Pentostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: pentostatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining pentostatin and cyclophosphamide with rituximab in treating patients who have chronic lymphocytic leukemia or lymphocytic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of pentostatin, cyclophosphamide, and rituximab, in terms of response rate, time to treatment failure, time to disease progression, durability of response, and overall survival, in patients with B-cell chronic lymphocytic leukemia or small B-cell lymphocytic lymphoma.
* Determine the safety of this regimen, in terms of acute, subacute, and chronic toxicity, in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy (no prior chemotherapy for chronic lymphocytic leukemia vs prior purine analog-based therapy [fludarabine or cladribine] but no alkylator therapy vs prior alkylator-based therapy [chlorambucil or cyclophosphamide] but no prior purine analog therapy vs prior therapy with alkylators and purine analogs, but not as combination therapy).

* First course: Patients receive rituximab IV over 1-4 hours on days 1-3 and pentostatin IV over 10-30 minutes and cyclophosphamide IV over 30-60 minutes on day 1.
* All subsequent courses: Patients receive rituximab IV over 60 minutes, pentostatin IV over 10-30 minutes, and cyclophosphamide IV over 30-60 minutes on day 1. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 5 years.

PROJECTED ACCRUAL: A total of 160-240 patients (40-60 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia (CLL) or small B-cell lymphocytic lymphoma (SLL) with the following:

  * Lymph node biopsy interpreted as SLL or consistent with CLL or all of the following:

    * Peripheral lymphocyte count greater than 5,000/mm^3 with small to moderate peripheral lymphocytes and no more than 55% prolymphocytes
    * Bone marrow aspirate containing at least 30% lymphoid cells
    * Immunophenotypic evaluation of peripheral blood lymphocytes demonstrating monoclonality of B lymphocytes with all of the following:

      * CD19 or CD20 coexpressed with CD5 antigen in the absence of other pan-T- cell markers (e.g., CD2 or CD3)
      * Expression of CD23 on CLL cells or Dim B-cell expression of kappa or lambda light chains
* Measurable disease with any of the following:

  * 1 or more lymph nodes at least 1.5 cm by CT scan
  * Splenomegaly by CT scan
  * Peripheral lymphocyte count greater than 5,000/mm3 with coexpression of CD5 and B-cell markers
  * Bone marrow aspirate with at least 30% lymphoid cells
* No mantle cell lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 2 years

Hematopoietic

* See Disease Characteristics
* No immune thrombocytopenia
* No hemolytic anemia

Hepatic

* Bilirubin no greater than 3 times upper limit of normal (ULN)
* SGOT no greater than 3 times ULN (unless due to hemolysis or CLL)
* No hepatitis

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* No cardiac dysfunction
* No New York Heart Association class III or IV heart disease
* No myocardial infarction within the past month

Other

* HIV negative
* No active acute or chronic infection
* No immunosuppressive diseases
* No autoimmune disorder
* No secondary malignancy that is projected to limit life expectancy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* No prior rituximab
* At least 4 weeks since prior biologic therapy

Chemotherapy

* At least 4 weeks since prior chemotherapy
* No prior combination chemotherapy and rituximab or other antibody therapy
* No prior combination chemotherapy comprising an alkylating agent and a purine nucleoside analog (i.e., cyclophosphamide or chlorambucil in combination with fludarabine, cladribine, or pentostatin)
* No prior pentostatin

Endocrine therapy

* At least 4 weeks since prior corticosteroids
* No concurrent supra-physiologic doses of corticosteroids

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* At least 4 weeks since prior major surgery

Other

* No concurrent immunosuppressive therapy (e.g., cyclosporine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Primary Completion 2004-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Cancer Center at Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States